CLINICAL TRIAL: NCT07182643
Title: An Exploratory Study of Biomarkers in the Endometrial Fluid, Tissue, and Follicular Fluid of Moderate/Severe Endometriosis Patients: a Prospective Study
Brief Title: Biomarkers in the Endometrial Fluid, Tissue, and Follicular Fluid of Moderate/Severe Endometriosis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2025-03224-01
Record Dates: First submitted 2025-09-09; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Endometriosis
Keywords: endometriosis; biomarkers; implantation; infertility; fertility
MeSH Terms: conditions — Endometriosis; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endometrial fluid, follicular fluid, endometrial biopsy, endometriosis lesions biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriosis: Moderate/severe endometriosis
  Interventions: Diagnostic Test: Endometrial fluid; Diagnostic Test: Endometrial biopsy; Diagnostic Test: Follicular fluid
- Controls: Healthy women undergoing oocyte pick up
  Interventions: Diagnostic Test: Endometrial fluid; Diagnostic Test: Endometrial biopsy

INTERVENTIONS:
Diagnostic Test: Endometrial fluid — Endometrial fluid collection in the day of OPU
Diagnostic Test: Endometrial biopsy — Endometrial biopsy on the OPU day, Pipelle
Diagnostic Test: Follicular fluid — Follicular fluid sampling on the OPU day
  Groups: Endometriosis

SUMMARY:
This study aims to explore biomarkers in the endometrial fluid and tissue of women with moderate to severe endometriosis, with a specific focus on those involved in pre-receptive endometrium and embryo implantation. This research has the potential to uncover diagnostic indicators of impaired pre-receptive endometrium, examine pathophysiological pathways, and identify future targets for therapeutic intervention. Ultimately, the findings may contribute to more personalized fertility treatments, offering new hope for women struggling with endometriosis-related infertility.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years old
* Diagnosed with moderate/severe endometriosis by ultrasound or laparoscopy (patient group)
* Regular menstrual cycles 28-35 days
* Speak English or Swedish and agree to participate in the study

Exclusion Criteria:

* Pregnancy or lactation in the last 3 months
* Uterine anomalies
* Pelvic inflammatory disease, endometritis, STD
* Gynaecological cancers or other malignancies in the patient's history
* Smoking (more than 10 cigarettes per day) or alcohol abuse
* Immunosuppressing medicines
* Major abdominal or pelvic surgery in the last 3 months
* A specific genetic disease that is diagnosed before PGT in women undergoing treatment

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We are going to recruit 30 patients who undergo fertility preservation or fertility treatment before endometriosis surgery in the Reproductive Medicine Clinic in Karolinska University Hospital. Our patients are diagnosed with stage III/IV endometriosis according to rASRM staging by using ultrasound. The control group will consist of 60 healthy women without endometriosis signs in the ultrasound who present to our clinic as oocyte donors or for fertility treatment because of male factor or pregenetic testing for genetic diseases of the partner
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Relative expression levels (e.g., fold change, normalized intensity, or concentration in pg/mL/ng/mL depending on biomarker assay) | 2 years
  Evaluation of the expression levels of selected biomarkers in endometrial fluid samples from patients with moderate to severe endometriosis compared to healthy controls.
Percentage of blastoids successfully implanted in vitro (% implantation rate) | 2 years
  Evaluation of the implantation efficiency of blastoids in vitro (endometrial organoids) under controlled laboratory conditions.

SECONDARY OUTCOMES:
Relative expression levels (e.g., concentration in pg/mL, ng/mL, or fold change depending on assay) | 2 years
  Assessment of biomarker expression levels in follicular fluid samples from follicles in different distances from endometriomas in patients with severe endometriosis.

CONTACTS AND LOCATIONS:
Overall Officials: Kenny Rodriguez-Wallberg, Professor, Principal Investigator — Onk/Pat Karolinska Institute
Locations (1):
- Karolinska Institute and Karolinska University Hospital Huddinge, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided